CLINICAL TRIAL: NCT03301337
Title: Amino-acid Uptake After Hydrolyzed Meat Protein Intake in Healthy Elderly
Brief Title: Amino-acid Uptake After Meat Protein Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: DC Ingredients (Unknown)
Responsible Party: Principal Investigator, Jakob Agergaard, Postdoc, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BBH 135
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Amino Acid Metabolism
Keywords: Amino acid uptake; Aging; Meat protein

STUDY DESIGN:
Intervention Model Description: Single-blindet randomized cross-over study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessor and investigator will be blindet. Participants cannot be blindet, as they will consume three different meat products, that we cannot mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrolyzed meat protein (Experimental): D5-phenylalanine intrinsically labelled hydrolyzed meat protein (0.6 g per kg lean body mass), which will be consumed together with a full meal.
  Interventions: Dietary Supplement: Meat protein absorption
- Minced Meat (Experimental): D5-phenylalanine intrinsically labelled hydrolyzed meat protein (0.6 g per kg lean body mass), which will be consumed together with a full meal.
  Interventions: Dietary Supplement: Meat protein absorption
- Beef (Experimental): D5-phenylalanine intrinsically labelled hydrolyzed meat protein (0.6 g per kg lean body mass), which will be consumed together with a full meal.
  Interventions: Dietary Supplement: Meat protein absorption

INTERVENTIONS:
Dietary Supplement: Meat protein absorption — Meat protein absorption when digested together with a full meal.

SUMMARY:
The purpose of the project is to provide evidence for the use of hydrolysed meat protein (HMP) as a protein supplement for elderly who has difficulty meeting the recommended daily protein intake.

The study will investigate how the meat protein derived amino acids (from either HMP, steak or minced meat) are absorbed and released into the blood circulation of elderly persons. Hereby, the study will explore the the anabolic potential of HMP compared with common meat products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Untrained

Exclusion Criteria:

* below 65 years of age
* BMI above 30
* Smokers
* Vegetarians
* Subjects with diabetes or other metabolic diseases
* Medical treatment affecting protein synthesis
* Gastro-intestinal problems, reduced liver or kidney function, elevated blood pressure, atherosclerosis
* More than 5 ours regular physical activity per week (except physical activity related to commuting)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
D5-phenylalanine appearance | 5 hours
  D5-phenylalanine appearance in the blood circulation after meal consumption

SECONDARY OUTCOMES:
Insulin concentration | 5 hours
  Insulin concentration in the blood circulation after meal consumption

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Agergaard, PhD, Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Denmark